CLINICAL TRIAL: NCT01821027
Title: A Open-Label, Single Sequence Study to Assess the Pharmacokinetics and Pharmacodynamics of Simvastatin Alone and of Simvastatin in Combination With JNJ-28431754 in Healthy Adult Subjects
Brief Title: A Study to Assess the Effects of Canagliflozin (JNJ-28431754) on the Pharmacokinetics, Pharmacodynamics, and Safety of Simvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015511; 28431754DIA1009 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Pharmacodynamics; Simvastatin (ZOCOR)
MeSH Terms: interventions — Simvastatin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canagliflozin + simvastatin (Experimental): Each volunteer will receive a single dose of simvastatin on Day 1, followed by canagliflozin (JNJ-28431754) once daily on Days 2 through 6. On Day 7 volunteers will receive a single dose of simvastatin in combination with a single dose of canagliflozin.
  Interventions: Drug: Simvastatin; Drug: Canagliflozin (JNJ-28431754)

INTERVENTIONS:
Drug: Simvastatin — One 40 mg tablet taken orally (by mouth) on Day 1 and Day 7.
  Other Names: Zocor
Drug: Canagliflozin (JNJ-28431754) — One 300 mg dose (ie, one 100 mg and one 200 mg over-encapsulated tablet) taken orally (by mouth) on Days 2 through Day 7.
  Other Names: JNJ-28431754

SUMMARY:
The purpose of this study is to determine how multiple doses of canagliflozin (JNJ-28431754) affect the pharmacokinetics (ie, how the body affects the drug) and pharmacodynamics (ie, how the drug affects the body) of a single dose of simvastatin.

DETAILED DESCRIPTION:
This study will be an open-label (all volunteers and study staff know the identity of the assigned treatment), single-center, fixed-sequence study (all volunteers receive the same medication on the same days and in the same order) to determine how multiple doses of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) affects the pharmacokinetics and pharmacodynamics of a single dose of simvastatin (a drug used to treat raised cholesterol). The study will consist of 3 phases: a screening phase, an open-label treatment phase, and an end-of-study (or follow-up) phase. During the open-label treatment phase, each volunteer will receive a single 40 mg dose of simvastatin on Day 1, followed by 300 mg of canagliflozin once daily on Days 2 through 6. On Day 7, volunteers will receive both simvastatin 40 mg and canagliflozin 300 mg. Each volunteer will participate in the study for approximately 32 days

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI) (weight in kg/height in m2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Volunteers must be non-smokers

Exclusion Criteria:

- History of, or current active illness, considered to be clinically significant by the Investigator, or any other illness that the Investigator considers should exclude the patient from the study, or that could interfere with the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of simvastatin | Up to Day 8
  Comparison of plasma concentrations of simvastatin following administration of a single dose of simvastatin alone or in combination with multiple doses of canagliflozin (JNJ-28431754). This will be used to determine whether there is a pharmacokinetic interaction between simvastatin and canagliflozin.
Plasma concentrations of the active beta-hydroxyacid metabolite of simvastatin | Up to Day 8
  Comparison of plasma concentrations of the active metabolite of simvastatin following administration of a single dose of simvastatin alone or in combination with multiple doses of canagliflozin (JNJ-28431754). This will be used to determine whether there is a pharmacokinetic interaction between simvastatin and canagliflozin.
Plasma concentrations of active 3-hydroxy-3-methyl-glutaryl-coenzyme A (HMG-CoA) reductase inhibitory activity | Up to Day 8
  Comparison of plasma HMG-CoA reductase inhibitory activity following administration of a single dose of simvastatin alone or in combination with multiple doses of canagliflozin (JNJ-28431754). This will be used to determine whether there is a pharmacodynamic interaction between simvastatin and canagliflozin. (Simvastatin lowers cholesterol by inhibiting the activity of the enzyme HMG-CoA reductase).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Murphy J, Skee D, Wajs E, Mamidi RN, Tian H, Vandebosch A, Wang SS, Verhaeghe T, Stieltjes H, Usiskin K. Effect of canagliflozin on the pharmacokinetics of glyburide, metformin, and simvastatin in healthy participants. Clin Pharmacol Drug Dev. 2015 May-Jun;4(3):226-36. doi: 10.1002/cpdd.166. Epub 2014 Oct 27. PMID 27140803